CLINICAL TRIAL: NCT05354323
Title: An Open-label, Phase I Multicenter, Clinical Trial of NECVAX-NEO1 in Addition to Anti-PD-1 or Anti-PD-L1 Monoclonal Antibody Checkpoint Inhibitor Monotherapy in Patients With Solid Tumors
Brief Title: NECVAX-NEO1 in Addition to Checkpoint Inhibitor in Patients With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NEC OncoImmunity AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NECVAX-NEO1-LT
Record Dates: First submitted 2022-04-19; First posted 2022-04-29 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NECVAX-NEO1 (Experimental): Personalized patient-individual oral DNA vaccine
  Interventions: Biological: NECVAX-NEO1

INTERVENTIONS:
Biological: NECVAX-NEO1 — Oral Ty21a based T-cell vaccination, personalized patient-individual NECVAX-NEO1 constructs containing a eukaryotic expression plasmid encoding for a series of selected neoantigen epitopes

SUMMARY:
NECVAX-NEO1 in addition to anti-PD-1 or anti-PD-L1 monoclonal antibody checkpoint inhibitor monotherapy in n=6 patients with solid tumors

DETAILED DESCRIPTION:
The trial is conducted as a multi-centre, open label, single-arm phase 1 first-in-human trial to evaluate NECVAX-NEO1, a personalized investigational oral cancer immunotherapeutic investigational medicinal product in n=6 patients with solid tumors under anti-PD-1 or anti-PD-L1 monoclonal checkpoint inhibitor monotherapy.

The trial has been designed to assess safety and tolerability of NECVAX-NEO1, at two dose levels as well as efficacy signals of NECVAX-NEO1 and immuno- and biomarkers in tumor tissue and blood samples pre- and post treatment.

The trial will include patients with a diagnosis of either non-small cell lung cancer (NSCLC), melanoma, urothelial cancer, renal cell cancer (RCC), or squamous cell cancer of head and neck (SCCHN). Neoantigen epitopes as patient-individual tumor-specific drug targets will be selected and identified by the NEC OncoImmunity proprietary machine-learning and artificial intelligence technology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to understand and follow instructions during the trial.
2. Patients able and willing to give written informed consent, signed and dated.
3. Male or female patients.
4. Patients aged 18 to 75 years old inclusive at the time of ICF signature.
5. Cancer patients with measurable disease according to RECIST 1.1, treated for at least three (3) months with an anti-PD-1 or anti-PDL1 checkpoint inhibitor as first- or second-line monotherapy, according to the Summary of Product Characteristics (SmPC) and national/institutional guidelines, for one of the following tumor types:

   1. non-small cell lung cancer, or
   2. cutaneous melanoma, or
   3. urothelial carcinoma, or
   4. renal cell carcinoma, or
   5. squamous cell cancer of head and neck.
6. Patients with SD or PR according to RECIST 1.1 at Screening
7. Patients with tumor or metastasis accessible for guided needle biopsy or resectable tumor in case of cutaneous melanoma when needle biopsy is not performed.
8. Patients with adequate bone marrow function, including:

   1. ANC ≥ 1.5 × 109/L; patients with documented benign cyclical neutropenia are allowed if white blood cell count is ≥ 1.5 × 10E9/L, with ANC ≥ 1.0 × 10E9/L, leukocytes ≥ 4.0 × 10E9/L, and lymphocytes ≥ 0.6 × 10E9/L;
   2. platelets ≥ 100 × 10E9/L;
   3. hemoglobin ≥ 9 g/dL (may have been transfused);
9. International Normalized Ratio (INR) < 1.5 × Upper Limit of Normal (ULN); patients treated with vitamin K antagonist are eligible if INR < 3.
10. Patients with adequate hepatic function at Screening, confirmed at Baseline, defined by

    1. total bilirubin level ≤ 1.5 × ULN; patients with documented Gilbert disease are allowed if total bilirubin ≤ 3 × ULN;
    2. aspartate aminotransferase (AST) level ≤ 2.5 × ULN, and alanine aminotransferase (ALT) level ≤ 2.5 × ULN, or, for patients with documented metastatic disease to the liver, AST and ALT levels ≤ 5 × ULN.
11. Patients with adequate renal function at Screening, confirmed at Baseline, defined by an estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula.
12. Patients must be able to undergo MRI or CT scan for tumor follow-up.
13. Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
14. Life expectancy of at least six (6) months according to the Investigator's judgement.

Exclusion Criteria:

Medical and surgical history, and diseases

1. History of any disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, based on the Investigator's judgement, provides a reasonable suspicion of a disease or condition that contraindicates the use of the IMP or that might affect the interpretation of the trial results or render the patient at high risk for treatment complications.
2. Brain metastasis.
3. Previously reported immune-related checkpoint inhibitor side effects of CTCAE Grade 3 or higher not having resolved to Grade 1 within six (6) weeks before inclusion.
4. Any significant co-morbidity which, according to the Investigator's judgement, makes patient compliance to trial conditions unlikely.
5. Previous malignant disease (other than the tumor disease for this trial) within the last five (5) years (except adequately treated non-melanoma skin cancers and carcinoma in situ of skin, bladder, cervix, colon/rectum, breast, or prostate) unless a complete remission without further recurrence was achieved at least two (2) years prior to Screening, and the patient is deemed to have been cured with no additional therapy required or anticipated to be required.
6. Prior organ transplantation, including allogeneic stem cell transplantation.
7. Congenital or any other immunodeficiency syndromes, or any active autoimmune disease that might deteriorate when receiving an immunostimulatory agent, except for:

   1. patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment, who are eligible.
   2. administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation), which is acceptable.
8. History of uncontrolled intercurrent illness, including but not limited to uncontrolled diabetes (e.g., hemoglobin A1c ≥ 8%);
9. Known prior hypersensitivity to the IMP or any component in its formulations or any other drug scheduled or likely to be given during the trial, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥ 3).
10. Persisting toxicity related to prior therapy (NCI CTCAE v5.0 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 AEs not constituting a safety risk based on Investigator's judgement are acceptable.
11. Other severe acute or chronic medical conditions, including immune colitis, inflammatory bowel disease, history of severe vomiting or diarrhea not having resolved to Grade 1 at Baseline, immune pneumonitis, pulmonary fibrosis, or psychiatric conditions including recent (within the last year) or active suicidal ideation or behavior, or laboratory abnormalities that may increase the risk associated with trial participation or trial treatment administration or may interfere with the interpretation of trial results and, in the judgement of the Investigator, would make the patient inappropriate for entry into this trial.
12. History of small intestine resection surgery or other major gastrointestinal surgery.
13. Active infection requiring systemic therapy.
14. Known history of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome or multi-drug resistant gram-negative bacteria.
15. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at Screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody Screening test positive).
16. Women of childbearing potential. Prior and concomitant medication
17. Live vaccines within 30 days prior to trial treatment.
18. Treatment in any other clinical trial within 30 days or within five (5) half-lives of any prior treatment, before Screening;
19. Any other condition or treatment that, in the opinion of the Investigator, might interfere with the trial, or current drug or substance abuse;
20. Chronic concurrent therapy within two (2) weeks before the trial treatment or expected therapy during the trial treatment period with:

    1. corticosteroids (except steroids up to equivalent of dexamethasone 4 mg daily dose).
    2. immunosuppressive agents.
    3. antibiotics.
    4. any other anticancer therapy or concurrent anticancer treatment, for example, cytoreductive therapy, radiotherapy [with the exception of palliative short course, limited field (ie, ≤ 10 fractions and ≤ 30% bone marrow involvement or per institutional standard) radiotherapy, which may be administered during the trial. However, IMP dosing must be suspended at least 14 days prior to the start of radiotherapy and must not be resumed until at least 14 days after the last radiotherapy fraction], immune therapy, or cytokine therapy, except for erythropoietin.

    Other
21. Inability to understand the Protocol requirements, instructions and trial-related restrictions, the nature, scope, and possible consequences of the trial.
22. Unlikely to comply with the Protocol requirements, instructions and trial-related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the trial.
23. Legal incapacity or limited legal capacity.
24. Any condition which results in an undue risk for the patient during the trial participation according to the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | 36 weeks
  AEs listed including system organ class, preferred term, severity, causality and other possibly relevant information. Frequency tables (including both patient and event counts) by System Organ Class (SOC) and preferred term (in number and percentage)

SECONDARY OUTCOMES:
Overall Response Rate ORR | 36 weeks
  ORR according to RECIST 1.1 with frequencies and percentages (in number and percentage)
Progression-Free Survival PFS | 36 weeks
  PFS measured from the date of enrolment to the date of first documentation of progression or death (from any cause), whichever occurs first (in days).
Time to Progression TTP | 36 weeks
  TTP measured from the date of enrolment to the date of first documentation of progression or death (from any cause), whichever occurs first, but deaths from other causes are censored at the date of death (in days)
Overall Survival OS | 36 weeks
  OS measured from the date of enrolment to the date of death resulting from any cause. Patients alive are censored at the time of last follow-up (in days).
Immune Response | 24 weeks
  ELISpot by descriptive analysis including changes from baseline at each post-baseline visit (in spot counts)

OTHER OUTCOMES:
Intratumoral T-cells | 24 weeks
  Tumor T-cell count at Week 24 compared to Baseline (in number of cells)
Intratumoral Tregs | 24 weeks
  Tumor Treg count at Week 24 compared to Baseline (in number of cells)

CONTACTS AND LOCATIONS:
Overall Officials: Elona Juozaityte, MD, Principal Investigator — Hospital of Lithuanian University of Health Sciences Kauno Klinikos
Locations (3):
- Lithuania (3):
  - Kaunas University Hospital, Kaunas
  - National Cancer Institute, Vilnius
  - Vilnius University Hospital Santaros Clinics, Vilnius

IPD SHARING:
Plan to Share IPD: Yes